CLINICAL TRIAL: NCT04581408
Title: Mutation-specific Therapy for the Long QT Syndrome
Acronym: MAST2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 26A804
Record Dates: First submitted 2020-09-27; First posted 2020-10-09 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Long QT Syndrome
Keywords: Long QT syndrome; Sudden cardiac death; Channelopathy; Gene-specific therapy; Life-threatening arrhythmias
MeSH Terms: conditions — Long QT Syndrome; Death, Sudden, Cardiac; Channelopathies | interventions — lumacaftor; ivacaftor; lumacaftor, ivacaftor drug combination

STUDY DESIGN:
Intervention Model Description: Open label, single arm, before vs after treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Orkambi (Experimental): Generic name: Lumacaftor/Ivacaftor
  Dosage form: tablet
  Dosage: each tablet contains 200 mg of Lumacaftor and 125 mg of Ivacaftor
  Frequency: two tablets twice a day.
  Interventions: Drug: Lumacaftor / Ivacaftor, Orkambi® Oral Tablet

INTERVENTIONS:
Drug: Lumacaftor / Ivacaftor, Orkambi® Oral Tablet — Total daily dose: 800 mg of Lumacaftor and 500 mg of Ivacaftor.
  Duration of treatment: according to the clinical conditions of the patient and based on the response to the drugs: up to a maximum of 7 days
  Other Names: Orkambi

SUMMARY:
Novel therapy for the Long QT Syndrome based on the mechanism of action of the disease-causing mutations

Long QT syndrome type 2 (LQT2) accounts for ~ 35% of all LQTS cases and is difficult to manage, as beta-blockers frequently fail to provide full protection. Most LQT2 patients (pts) have a Class 2 mutation, which implies defective "trafficking".

Lumacaftor (LUM) is a drug developed and currently indicated for the treatment of cystic fibrosis (CF) in patients homozygous for the F508del mutation in the CFTR gene. LUM corrects protein folding and trafficking defects of mutant and misfolded CFTR channels, restoring their cell surface expression. The investigators recently demonstrated that LUM can rescue in vitro the LQTS phenotype observed in human induced pluripotent stem cell- derived cardiomyocytes (hiPSC-CMs) from pts with LQT2 Class 2 mutations (PMID: 29020304) and in these same two patients Orkambi administrated for 7 days at the same dosage approved for cystic fibrosis showed to reduce their QTc (PMID: 30753398).

With the present phase II clinical trial (MAST2) the investigators will enroll 20 LQT2 patients (see inclusion and exclusion criteria) and they will test in vivo the efficacy of Orkambi in shortening their QTc. Patients will be admitted to hospital for a maximum of 7 days (minimum in-hospital stay based on evidence of QTc shortening). Orkambi will be administered at the dose approved for cystic fibrosis and during the entire period continuous ECG monitoring through both telemetry and 12-lead 24-hr Holter monitoring will be performed and QTc length and morphology will be analyzed.

DETAILED DESCRIPTION:
The congenital Long QT Syndrome (LQTS) is a life-threatening condition characterized by a prolonged QT interval on the electrocardiogram, and an increased risk of life-threating arrhythmias in otherwise healthy individuals. Typically, the heart is structurally normal and the electric abnormality present in these patients is due to mutations in genes encoding ion channel subunits or proteins modulating ion-channel function. The investigators will specifically study the LQT2 variant which is the second most common form of LQTS (30-35% of all LQTS cases), a rare condition present in approximately 1 in 7.500-8.000 live births characterized by loss-of-function mutations in the KCNH2 gene (hERG) which result in a reduction of the potassium current IKr, pivotal for ventricular repolarization. Four different mutation classes define the molecular mechanisms impairing hERG. Among these, almost 50% are class 2 mutations that determine hERG trafficking defects, with the consequent lack of expression of these essential ion channels on the cardiomyocyte membrane.

According to clinical severity current therapies for LQT2 include β-blockers, left cardiac sympathetic denervation and an implantable cardioverter defibrillator (ICD). However, ICD implantation, is not devoid of complications and often, the pain and fear associated with ICD shocks lead to electrical storms with multiple recurrent shocks. Furthermore, there are concerns about the long-term impact of implanting an ICD in young LQTS patients, likely to live another 7 to 8 decades after initial device implantation and who would be subjected to multiple procedures for generator replacement and lead revisions/extractions with frequent complications. There is a clear and unmet need for additional therapeutic strategies and implementation of gene-specific therapy could represent a quite important step for improving the clinical management of these pts.

Lumacaftor (LUM) is a drug developed and currently indicated for the treatment of cystic fibrosis (CF) in patients aged 12 years and older who are homozygous for the F508del mutation in the CFTR gene. By acting as a chaperone, LUM corrects protein folding and trafficking defects of mutant and misfolded CFTR channels, restoring their cell surface expression. In its commercial formulation - brand name Orkambi - it is combined with ivacaftor (IVA), an enhancer of the CFTR protein function. The recommended dose is two tablets (each tablet containing LUM 200 mg/ IVA 125 mg) taken orally every 12 hours for a total daily dose of LUM 800 mg/ IVA 500 mg.

The investigators recently demonstrated that LUM can rescue in vitro the LQTS phenotype observed in human induced pluripotent stem cell- derived cardiomyocytes (hiPSC-CMs) from patients with LQT2 Class 2 mutations (PMID: 29020304) and in these same two patients Orkambi administrated for 7 days at the same dosage approved for cystic fibrosis showed to reduce their QTc (PMID: 30753398).

With the present phase II clinical trial (MAST2) 20 LQT2 patients will be enrolled (see inclusion and exclusion criteria). Patients will be admitted to hospital for a maximum of 7 days (minimum in-hospital stay based on evidence of QTc shortening) while beta-blocker therapy will continue at the current dose. Orkambi will be administered at the dose approved for cystic fibrosis [Orkambi (Lumacaftor 200 mg/Ivacaftor 125 mg) 2 tablets twice a day for a total daily dose of 800 mg of Lumacaftor and 500 mg of Ivacaftor] and blood exams will be performed at day 1, 3, 5 and 7. During the entire period continuous ECG monitoring through both telemetry and 12-lead 24-hr Holter monitoring will be performed and QTc length and morphology will be analysed. Independently of the result the patient will be discharged without Orkambi as a chronic therapy. Therefore, the drug will be administered orally for a maximum of 7 days.

In case of side effects a reduction of the dose will be considered and according to the specific problem the possibility of an interruption will be evaluated. Furthermore, as an additional "stopping rule" the patient can freely decide to withdraw from the study in any moment even during the Hospitalization phase.

Compliance will be strictly monitored as the drug will be assumed in Hospital in front of the nurse twice a day for the maximum of 7 days. Placebo will not be used.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent: it is requested that the partipants understand the nature of the study and can give their voluntary conset after being fully informed, after having received satisfying replies to their questions regarding the study, and all the authorizations according to local requirements. The informed consent form was previously approved by the local Ethics Committee and will have to be dated and signed before enrollment in the study.
* Age and gender: participants of both the male and female sex aged between 18 and 65 years will be included
* Mutations: the study will enrol patients with LQT2, i.e., with pathogenic mutations on the KCNH2 gene, that present such functional characterization that classifies them as class II mutations, namely mutations that cause a trafficking defect. This characterization includes, but is not limited to, patch clamp data in single cells, immunofluorescence data, positive reactions to drugs that correct the trafficking defect in vitro.
* Consent of the patient to not participate in any other clinical study during the entire period of participation in the present study
* Women with child-bearing potential (pre-menopausal women, less than two years after start of menopause and women who are not surgically sterile) must use a highly effective contraceptive method from 30 days before enrollment in the study until 28 days after the last administration of study drug. It is specified that the sole use of hormonal contraception, both oral, injectable, transdermic and implantable cannot be considered an effective contraceptive method. Orkambi (Lumacaftor/ivacaftor) may reduce the exposure to the hormonal contraceptives and possibly cause their ineffectiveness. Male patients with a female partner with child-bearing potential must use 2 forms of contraception (one of which should be a double-barrier method) from enrolment in the study until 28 days after the last administration of study drug. Highly effective contraceptive methods are: i) abstinence, ii) surgical sterilization (=6 months postsurgery), iii) intrauterine device or intrauterine system, iv) oral contraceptives combined with a barrier method, v) double-barrier method (e.g., male condom or diaphragm with vaginal spermicides).

Exclusion Criteria:

* Absence of one or more of the preceeding inclusion criteria
* Hypersensitivity to the active substance (to one or both active substances) or to one of the excipients.
* Pregnancy (established before enrollment by positive urine pregnancy test in potentially fertile women) or breastfeeding
* Participation in a clinical study in which an experimental drugs has been administered less than 30 days or less than 5 half-lives before the present study drug
* Any clinical condition that in the opinion of the investigator causes the patients not to be suitable for the study and/or that may involve an unreasonable/significant risk for the participants, thereby changing the interpretation of that data and affecting the continuation of the study
* Other important cardiac diseases and in particular: cardiomyopathies and myocarditis, pericardial diseases, other associated channelopathies, ischemic heart disease, heart failure, pulmonary heart disease, severe valuvulopathies, rhythm alterations such as atrial fibrillation or atrial flutter, complete right or left bundle branch block, advanced atrio-ventricular blocks, uncontrolled arterial hypertension on beta-blocker therapy
* Significant extracardiac diseases and in particular:

  * renal failure. In accordance with the SmPC, patients with severe (estimated GFR <30 mL/min/1.73 m2) and moderate (estimated GFR 30-60 mL/min/1.73 m2) renal impairment at screening are excluded
  * impairment of liver function. In accordance with the SmPC, patients with severe (Child-Pugh Class C) and moderate (Child-Pugh Classe B) liver function impairment are excluded
  * important diseases of the respiratory system and in particular: any pulmonitis, obstructive bronchopulmonary disease with FEV1 <80%, asthmatic bronchitis, infiltrative lung disease, lung emboly, pulmonary hypertension, idiopathic pulmonary fibrosis, pneumothorax, neoplasms of lungs and pleura
  * important neurological diseases and in particular: epilepsy, cerebral hemorrhage, stroke, multiple sclerosis, cerebral tumours, cerebral or spinal traumas, Parkinson's disease, cognitive deterioration and Alzheimer's disease
* Chronic use of therapies other than beta-blocker treatment and intake of any potassium/magnesium supplement that the patient may use chronically or intermittently (oral contraceptives are allowed, but must be interrupted during the study).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
QT interval | 3 to 7 days after start of treatment
  Change in QT interval after drug treatment

CONTACTS AND LOCATIONS:
Overall Officials: Lia Crotti, MD, Principal Investigator — Istituto Auxologico Italiano; Peter J Schwartz, MD, Study Director — Istituto Auxologico Italiano
Locations (1):
- Istituto Auxologico Italiano, Ospedale San Luca, Milan, Italy

IPD SHARING:
Plan to Share IPD: No